CLINICAL TRIAL: NCT04085939
Title: Referral to Pharmacists - Ambulance Clinician Experience Survey
Acronym: REPLACES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yorkshire Ambulance Service NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: YASRD123
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pharmacist-Patient Relations; Fall Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online survey — Anonymous survey using the online survey tool, JotForm

SUMMARY:
Falls in people aged 65 years and over are a common reason for calling the emergency ambulance service. Falls can be serious, with about 1 in 20 people having to be taken to hospital because they have been injured. Thankfully, in more than 4 out of 10 cases, people are not seriously injured and can be left at home. However, it is important that the reason for the fall is found and future falls are prevented where possible.

Yorkshire Ambulance Service can already make a referral to another local service to get specialist practical help for falls prevention when people are left at home after a fall. Research has shown that the safe use of medicines can prevent future falls, but that did not form. Now a new service has been set up for Yorkshire Ambulance Service to refer patients to the Leeds General Practice (GP) Confederation. A pharmacist working in the patients GP surgery will undertake a review of the patient's use of their medicines.

However, it is unknown how ambulance staff identify patients who may be at risk of future falls due to medicines being taken or issues with medicines management at home. This data is not currently collected in any ambulance patient records. It is also not known what their current practice is when a patient who is not managing their medicines well is identified. A literature search has revealed no papers on this topic. This research survey seeks to understand how ambulance clinicians identify and assist patients who are having difficulty in managing their medicines. Therefore, the results of this study are likely to provide new knowledge which will be generalisable to United Kingdom (UK) ambulance service practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical staff working operationally, providing frontline ambulance care in Yorkshire Ambulance Service National Health Service (NHS) Trust during the PREFACES project (24th May, 2019 to 31st May 2020)

Exclusion Criteria:

* Clinical staff NOT working operationally, providing frontline ambulance care in Yorkshire Ambulance Service NHS Trust
* Non-clinical staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical staff working operationally, providing frontline ambulance care in Yorkshire Ambulance Service NHS Trust during the PREFACES project (24th May, 2019 to 31st May 2020)
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Weighted average of factors that identify patients having difficulty managing their medicines, ranked in order of importance by ambulance clinicians | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Yorkshire Ambulance Service NHS Trust, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No